CLINICAL TRIAL: NCT00824421
Title: A Phase 2B Multicenter, Randomized, Double-Blind, Comparative Trial Of UK-453,061, In Combination With Tenofovir Df And Emtricitabine Versus Efavirenz In Combination With Tenofovir DF And Emtricitabine For The Treatment Of Antiretroviral-Naive HIV-1 Infected Subjects
Brief Title: A Study Of Different Doses Of UK-453, 061 Plus Truvada Compared To Efavirenz Plus Truvada In Patients Who Have Not Been Previously Treated For HIV-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5271015
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2011-11

CONDITIONS: HIV-1
Keywords: HIV-1. Treatment Naive; HIV Infections; treatment naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- UK- 453,061 Dose One (Experimental): UK 453,061 Dose One plus Truvada
  Interventions: Drug: UK-453, 061
- UK-453,061 Dose Two (Experimental): UK 453,061 Dose Two plus Truvada
  Interventions: Drug: UK-453, 061
- Efavirenz + Truvada (Active Comparator): Efavirenz + Truvada
  Interventions: Drug: EFV +TVA

INTERVENTIONS:
Drug: UK-453, 061 — UK-453,061 500 mg tablets PO QD + Tenofovir DF 300 mg/Emtricitabine 200 mg tablets PO QD.
  Arms: UK- 453,061 Dose One
Drug: UK-453, 061 — UK-453,061 750 mg tablets PO QD + Tenofovir DF 300 mg/Emtricitabine 200 mg tablets PO QD.
  Arms: UK-453,061 Dose Two
Drug: EFV +TVA — Efavirenz 600 mg tablets PO QD + Tenofovir DF 300 mg/Emtricitabine 200 tablets mg PO QD.
  Arms: Efavirenz + Truvada

SUMMARY:
This is a 96 week study to determine if UK- 453,061 in combination with Truvada is as efficacious, safe and tolerable as efavirenz in combination with Truvada in HIV-1 infected patients who have not been previously treated with antiretroviral drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age available for a follow-up period of at least 96 weeks.
* HIV 1 RNA viral load of greater then 1,000 copies/mL
* Negative urine pregnancy test.

Exclusion Criteria:

* Suspected or documented active, untreated HIV-1 related opportunist infection or other condition requiring acute therapy at the time of randomization.
* Subjects with acute Hepatitis B and/or C within 30 days of randomization.
* Absolute CD4 count <200 cells/mm3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- Pfizer Investigational Site, Buenos Aires, Argentina
- Australia (2):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Melbourne, Victoria
- Canada (2):
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Italy (2):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Torino
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico
- Poland (4):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Warsaw
- South Africa (7):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Soweto, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Namakgale, Limpopo
  - Pfizer Investigational Site, Cape Town, Western Cape
  - Pfizer Investigational Site, Pretoria
- Switzerland (3):
  - Pfizer Investigational Site, Ch-8091 Zurich
  - Pfizer Investigational Site, Lugano
  - Pfizer Investigational Site, Sankt Gallen
- United Kingdom (4):
  - Pfizer Investigational Site, Crumpsall, Greater Manchester
  - Pfizer Investigational Site, Brighton
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271015&StudyName=A%20Study%20Of%20Different%20Doses%20Of%20UK-453%2C%20061%20Plus%20Truvada%20Compared%20To%20Efavirenz%20Plus%20Truvada%20In%20Patients%20Who%20Have%20Not%20Been%20Previously

RESULTS

PARTICIPANT FLOW:
Groups:
- Lersivirine 500 mg: Two lersivirine 250 milligram (mg) tablets (equivalent to lersivirine 500 mg), a placebo tablet matched to lersivirine and a placebo tablet matched to efavirenz orally once daily along with tenofovir disoproxil fumarate (DF) 300 mg tablet and emtricitabine 200 mg tablet orally once daily, in the evening up to 96 weeks. Participants enrolled in pharmacokinetic (PK) substudy switched to lersivirine morning dosing regimen, received 2 Lersivirine 250 mg tablets, a placebo tablet matched to lersivirine orally once daily in the morning for 7 days prior to Week 4, and in the morning and evening on 1 day following Week 4. A placebo tablet matched to efavirenz, tenofovir DF 300 mg tablet and emtricitabine 200 mg tablet were continued in the evening in PK substudy. Evening dosing was continued for the remainder of the study up to Week 96.
- Lersivirine 750 mg: Three Lersivirine 250 mg tablets (equivalent to lersivirine 750 mg) and a placebo tablet matched to efavirenz orally once daily along with tenofovir DF 300 mg and emtricitabine 200 mg tablet orally once daily, in the evening up to 96 weeks. Participants enrolled in PK substudy switched to morning dosing regimen, received 3 Lersivirine 250 mg tablets orally once daily in the morning for 7 days prior to Week 4, and in the morning and evening on 1 day following Week 4. A placebo tablet matched to efavirenz, tenofovir DF 300 mg tablet and emtricitabine 200 mg tablet were continued in the evening in PK substudy. Evening dosing was continued for the remainder of the study up to Week 96.
- Efavirenz 600 mg: Three placebo tablets matched to lersivirine, efavirenz 600 mg tablet orally once daily along with tenofovir DF 300 mg and emtricitabine 200 mg tablet orally once daily, in the evening up to 96 weeks. Participants enrolled in PK substudy switched to morning dosing regimen, received 3 placebo tablets matched to lersivirine and efavirenz 600 mg tablet orally once daily in the morning for 7 days prior to Week 4, and in the morning and evening on 1 day following Week 4. Efavirenz 600 mg tablet, tenofovir DF 300 mg tablet and emtricitabine 200 mg tablet were continued in the evening in PK substudy. Evening dosing was continued for the remainder of the study up to Week 96.
Period: Overall Study
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Started | 66 | 66 | 63
Treated | 65 | 65 | 63
Completed | 49 | 44 | 49
Not Completed | 17 | 22 | 14
Not completed — Adverse Event | 6 | 6 | 6
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 5 | 7 | 4
Not completed — Lost to Follow-up | 2 | 3 | 0
Not completed — Pregnancy | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 3
Not completed — Randomized but not Treated | 1 | 1 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who had received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg | Total
Number analyzed (Participants) | 65 | 65 | 63 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.0) | 35.7 (8.2) | 36.3 (8.7) | 36.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 17 | 52
  Male | 49 | 46 | 46 | 141

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Less Than 50 Copies Per Milliliter (Copies/mL) of Human Immunodeficiency Virus Type 1 Ribonucleic Acid (HIV-1 RNA) at Week 48
Description: Plasma HIV-1 RNA level was determined by validated Roche Amplicor HIV-1 Monitor standard assay.
Time Frame: Week 48
Population: ITT population included all randomized participants who received at least 1 dose of study medication. Participants who had been discontinued from the study, were lost to follow-up, or had missing HIV-1 RNA level data at a visit were considered to have HIV-1 RNA levels >=50 copies/mL and were referred to as non-completer = failure.
Measure: Number; unit: percentage of participants
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 65 | 65 | 63
percentage of participants | 78.5 | 78.5 | 85.7

2. Secondary Outcome: Percentage of Participants With Less Than 50 Copies/mL of HIV-1 RNA at Week 24 and 96
Description: Plasma HIV-1 RNA level was determined by validated Roche Amplicor HIV-1 Monitor standard assay.
Time Frame: Week 24, 96
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 65 | 65 | 63
percentage of participants
  Week 24 | 83.1 | 83.1 | 87.3
  Week 96 | 70.8 | 67.7 | 77.8

3. Secondary Outcome: Percentage of Participants With Less Than 400 Copies/mL of HIV-1 RNA at Week 24, 48 and 96
Description: Plasma HIV-1 RNA level was determined by validated Roche Amplicor HIV-1 Monitor standard assay.
Time Frame: Week 24, 48, 96
Population: ITT population included all randomized participants who received at least 1 dose of study medication. Participants who had been discontinued from the study, were lost to follow-up, or had missing HIV-1 RNA level data at a visit were considered to have HIV-1 RNA levels >=400 copies/mL and were referred to as non-completer = failure.
Measure: Number; unit: percentage of participants
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 65 | 65 | 63
percentage of participants
  Week 24 | 84.6 | 87.7 | 90.5
  Week 48 | 81.5 | 80.0 | 85.7
  Week 96 | 73.8 | 67.7 | 77.8

4. Secondary Outcome: Change From Baseline in Log 10 Transformed HIV-1 RNA Levels at Week 24, 48 and 96
Description: For the log 10 scale, all the HIV-1 RNA levels were log 10 transformed prior to the average calculations. Baseline value was calculated as the average of all the measurements collected prior to and including Day 1 pre-dose.
Time Frame: Baseline, Week 24, 48, 96
Population: ITT population. Participant discontinued before a visit of interest: value imputed as zero; not discontinued but observation is missing: Last observation carried forward (LOCF) imputation used; missing baseline or no HIV-1 RNA level assessment: value imputed as zero.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 65 | 65 | 63
log 10 copies/mL
  Baseline | 4.62 (0.61) | 4.69 (0.66) | 4.66 (0.62)
  Change at Week 24 | -2.44 (1.19) | -2.63 (1.11) | -2.68 (1.05)
  Change at Week 48 | -2.36 (1.26) | -2.34 (1.33) | -2.52 (1.17)
  Change at Week 96 | -2.19 (1.38) | -1.98 (1.48) | -2.27 (1.34)

5. Secondary Outcome: Time-Averaged Difference (TAD) in Log 10 Transformed HIV-1 RNA Levels at Week 24, 48 and 96
Description: TAD was calculated as area under the curve of HIV-1 RNA levels (log10 copies/mL) from baseline to the time point of interest divided by time period in weeks minus baseline HIV-1 RNA level (log10 copies/mL). Baseline value was calculated as the average of all the measurements collected prior to and including Day 1 pre-dose.
Time Frame: Baseline up to Week 24, 48, 96
Population: ITT population. Participant discontinued before a visit of interest: value imputed as zero; not discontinued but observation was missing: value calculated to the last non-missing timepoint; not discontinued and missing values between baseline and visit: ignore missing values; missing baseline or no HIV-1 RNA level assessment: value imputed as zero.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 65 | 65 | 63
log10 copies/mL
  Week 24 | -2.17 (0.99) | -2.30 (0.94) | -2.40 (0.89)
  Week 48 | -2.23 (1.17) | -2.24 (1.19) | -2.39 (1.09)
  Week 96 | -2.16 (1.33) | -1.92 (1.43) | -2.21 (1.29)

6. Secondary Outcome: Percentage of Participants With Response as Determined Using the Time-to Loss of Virologic Response (TLOVR50) Algorithm at Week 24, 48 and 96
Description: TLOVR50 response is compliment to TLOVR50 failure. TLOVR50 failure based on observed HIV-1 RNA levels and failure events (death; permanent discontinuation of drug; lost to follow-up; met treatment failure [TF] criteria). TF: an increase to at least 3 times baseline plasma HIV-1 RNA level at Week 2 or thereafter; failure to achieve HIV-1 RNA level <50 copies/mL at Week 24; starting at Week 2, an increase in HIV-1 RNA level to detectable levels (>50 copies/mL). TF criteria's defined above were confirmed by second measurement at least 14 days after first. In 'TLOVR50', '50' denotes the lower limit of quantification (LLOQ) of assay (which is 50 copies/mL). Baseline value was calculated as the average of all the measurements collected prior to and including Day 1 pre-dose.
Time Frame: Week 24, 48, 96
Population: ITT population included all randomized participants who received at least 1 dose of study medication. Missing value was imputed per the TLOVR algorithm.
Measure: Number; unit: percentage of participants
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 65 | 65 | 63
percentage of participants
  Week 24 | 83.1 | 83.1 | 87.3
  Week 48 | 78.5 | 78.5 | 85.7
  Week 96 | 67.7 | 67.7 | 76.2

7. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD4+) Absolute Cell Count at Week 24, 48 and 96
Description: Baseline value was calculated as the average of all the measurements collected prior to and including Day 1 pre-dose.
Time Frame: Baseline, Week 24, 48, 96
Population: ITT population included all randomized participants who received at least 1 dose of study medication. LOCF method was used to impute missing values. No or zero change from baseline was imputed for participants with missing baseline or no CD4+ count available on treatment.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/mcL)
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 65 | 65 | 63
cells per microliter (cells/mcL)
  Baseline | 349 (120) | 352 (154) | 319 (80)
  Change at Week 24 | 146 (164) | 167 (127) | 139 (104)
  Change at Week 48 | 191 (206) | 195 (130) | 188 (117)
  Change at Week 96 | 215 (194) | 231 (187) | 221 (144)

8. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD4+) Percentage Cell Count at Week 24, 48 and 96
Description: Baseline value was calculated as the average of all the measurements collected prior to and including Day 1 pre-dose.
Time Frame: Baseline, Week 24, 48, 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of total lymphocytes
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 65 | 65 | 63
percentage of total lymphocytes
  Baseline | 19.9 (6.6) | 20.0 (6.7) | 19.5 (5.4)
  Change at Week 24 | 6.0 (4.1) | 7.5 (3.7) | 7.3 (4.7)
  Change at Week 48 | 8.3 (5.0) | 9.9 (4.3) | 8.7 (4.9)
  Change at Week 96 | 10.1 (6.4) | 12.1 (6.5) | 11.1 (6.0)

9. Secondary Outcome: Number of Participants With NRTI and NNRTI Resistance-Associated Mutations (RAMs) at Time of Treatment Failure Through Week 24, 48 and 96
Description: Phenotypic resistance and genotypic resistance was assessed for all participants at Day 1 predose, and was evaluated for nucleotide reverse transcriptase inhibitors (NRTIs), and non-NRTIs (NNRTIs) resistance-associated mutations at time of treatment failure using Monogram GenoSeq and/or PhenoSenseGT assays. This was then repeated for all participants with HIV-1 viral load more than 500 copies/mL at treatment failure, up to Week 96.
Time Frame: Day 1 (pre-dose) through Week 24, 48, 96
Population: Virology analysis set (TLOVR50 failures) included all participants who meet the TLOVR50 failure definition. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable for this measure at specified time point for each group, respectively.
Measure: Number; unit: participants
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 5 | 8 | 6
participants
  Week 24 (n=3, 4, 2) | 3 | 0 | 1
  Week 48 (n=4, 3, 3) | 3 | 1 | 1
  Week 96 (n= 5, 8, 6) | 3 | 1 | 1

10. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory analysis included hematology, blood chemistry, serum and urine pregnancy test, hepatitis testing and urinalysis. Laboratory values that met the criteria of the Division of Acquired Immuno Deficiency Syndrome (DAIDS) grade 1 (mild, symptoms causing no or minimal interference with usual social and functional activities) or greater were considered as abnormal.
Time Frame: Baseline up to Week 96 or early termination
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 64 | 65 | 63
participants | 59 | 58 | 57

11. Secondary Outcome: Population Pharmacokinetic (PK) of Lersivirine
Description: Data for this outcome measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the participant flow and baseline characteristics modules.
Time Frame: Week 2, 4, 8, 12, 16, 24, 32, 40, 48
Reporting Status: Not Posted

12. Secondary Outcome: Lersivirine Success Percentage With Reference to Median Minimum Observed Plasma Concentration (Cmin)
Description: Simple quartile exposure analysis of success rate (viral load <50 copies/mL) versus median Cmin assesses the exposure response relationship. Percentage of participants with HIV-1 RNA level <50 copies/mL at median Cmin quartile were planned to be reported.
Time Frame: Week 2, 4, 8, 12, 16, 24, 32, 40, 48
Population: Due to the sparsity of the data, it was deemed that the interpretation of the pharmacokinetic/pharmacodynamic (PK/PD) results would be questionable, thus data was not analyzed.
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) of Lersivirine
Description: AUC (0-24)= Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post-dose (0-24). Only participants from Lersivirine treatment arms were planned to be analyzed for Pharmacokinetic (PK) sub-study.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 24 hours (hrs) post-dose on Week 4
Population: Pharmacokinetic sub-study analysis set (PKSSAS) included all randomized Lersivirine participants who consented to participate in the PK sub-study, received the study medication on the day of the PK sub-study and had sufficient PK data for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- Lersivirine 500 mg: Participants enrolled in PK substudy received 2 Lersivirine 250 mg tablets and a placebo tablet matched to lersivirine orally once daily in the morning for 7 days prior to Week 4, and in the morning and evening on 1 day following Week 4. A placebo tablet matched to efavirenz, tenofovir DF 300 mg tablet and emtricitabine 200 mg tablet orally once daily were continued in the evening in PK substudy.
- Lersivirine 750 mg: Participants enrolled in PK substudy received 3 Lersivirine 250 mg tablets orally once daily in the morning for 7 days prior to Week 4, and in the morning and evening on 1 day following Week 4. A placebo tablet matched to efavirenz, tenofovir DF 300 mg tablet and emtricitabine 200 mg tablet orally once daily were continued in the evening in PK substudy.
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg
Number analyzed (Participants) | 7 | 6
nanogram*hour/milliliter (ng*hr/mL) | 6002 (30) | 8677 (21)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lersivirine
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 24 hrs post-dose on Week 4
Population: PKSSAS included all randomized Lersivirine participants who consented to participate in the PK sub-study, received the study medication on the day of the PK sub-study and had sufficient PK data for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg
Number analyzed (Participants) | 7 | 6
ng/mL | 1056 (41) | 1354 (31)

15. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Lersivirine
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 24 hrs post-dose on Week 4
Population: as for outcome 14
Measure: Median (Full Range); unit: hr
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg
Number analyzed (Participants) | 7 | 6
hr | 1.00 [0.483 to 2.00] | 2.00 [0.500 to 8.00]

16. Secondary Outcome: Plasma Concentration of Lersivirine at 24 Hour
Description: The observed plasma concentration at 24 hours post-dose (C 24h).
Time Frame: 24 hrs post-dose on Week 4
Population: PKSSAS included all randomized Lersivirine participants who further consented to participate in the PK sub-study, received the study medication on the day of the PK sub-study and had sufficient PK data for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg
Number analyzed (Participants) | 7 | 6
ng/mL | 49.56 (73) | 57.70 (34)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | Lersivirine 500 mg | Lersivirine 750 mg | Efavirenz 600 mg
Serious Adverse Events (participants affected / at risk) | 6/65 | 7/65 | 6/63
Other Adverse Events (participants affected / at risk) | 51/65 | 58/65 | 59/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lersivirine 500 mg (N=65) | Lersivirine 750 mg (N=65) | Efavirenz 600 mg (N=63)
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0 | 0
Syphilis (Infections and infestations) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Renal papillary necrosis (Renal and urinary disorders) | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lersivirine 500 mg (N=65) | Lersivirine 750 mg (N=65) | Efavirenz 600 mg (N=63)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 1 | 5
Chalazion (Eye disorders) | 0 | 0 | 2
Conjunctivitis (Eye disorders) | 3 | 5 | 2
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 1 | 0 | 0
Pterygium (Eye disorders) | 0 | 1 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 8 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2 | 1
Breath odour (Gastrointestinal disorders) | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 12 | 14
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 2
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 16 | 28 | 8
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1
Palatal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Palatal oedema (Gastrointestinal disorders) | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0
Poor dental condition (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 12 | 11
Asthenia (General disorders) | 2 | 2 | 4
Chest pain (General disorders) | 0 | 3 | 3
Cyst (General disorders) | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 4 | 3
Feeling abnormal (General disorders) | 0 | 0 | 2
Feeling drunk (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 3 | 5 | 2
Irritability (General disorders) | 2 | 1 | 1
Malaise (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 0
Pelvic mass (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0
House dust allergy (Immune system disorders) | 0 | 0 | 1
Immune reconstitution syndrome (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Balanitis candida (Infections and infestations) | 1 | 0 | 0
Body tinea (Infections and infestations) | 0 | 2 | 1
Borrelia infection (Infections and infestations) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 4 | 9 | 5
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Chlamydial infection (Infections and infestations) | 2 | 1 | 1
Conjunctivitis viral (Infections and infestations) | 1 | 0 | 0
Dysentery (Infections and infestations) | 0 | 0 | 1
Eyelid infection (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 2 | 2 | 2
Fungal skin infection (Infections and infestations) | 0 | 1 | 1
Furuncle (Infections and infestations) | 1 | 1 | 1
Gastroenteritis (Infections and infestations) | 5 | 5 | 5
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 2
Gonorrhoea (Infections and infestations) | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Herpes dermatitis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 4 | 0
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 1 | 0 | 0
Infected bites (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 5 | 7 | 8
Kaposi's varicelliform eruption (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 3 | 3
Molluscum contagiosum (Infections and infestations) | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 3 | 4
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 2 | 2
Oral hairy leukoplakia (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 2 | 2
Orchitis (Infections and infestations) | 0 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 2
Otitis media (Infections and infestations) | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 1
Parasitic gastroenteritis (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 1
Penile abscess (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 2 | 8
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 2 | 1
Rhinitis (Infections and infestations) | 3 | 1 | 2
Sinusitis (Infections and infestations) | 4 | 2 | 1
Skin candida (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 0
Syphilis (Infections and infestations) | 6 | 1 | 3
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 4 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 2 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 10 | 13 | 14
Urethritis (Infections and infestations) | 0 | 1 | 2
Urethritis chlamydial (Infections and infestations) | 1 | 0 | 0
Urethritis gonococcal (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 3
Vaginal infection (Infections and infestations) | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 4
Blood amylase increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 4
Blood creatinine increased (Investigations) | 2 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 2 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 2
Protein urine present (Investigations) | 1 | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 1 | 0
Vestibular function test (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 1 | 5
Weight increased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0
White blood cells urine (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Hand deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Areflexia (Nervous system disorders) | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 2 | 3
Dizziness (Nervous system disorders) | 5 | 5 | 15
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 3 | 1
Headache (Nervous system disorders) | 19 | 14 | 11
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 1
Somnolence (Nervous system disorders) | 3 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 2 | 1
Abnormal dreams (Psychiatric disorders) | 5 | 5 | 12
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 5 | 5
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 2 | 1
Depression (Psychiatric disorders) | 3 | 2 | 3
Disturbance in sexual arousal (Psychiatric disorders) | 0 | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 0 | 1
Grief reaction (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 7 | 9 | 8
Libido decreased (Psychiatric disorders) | 3 | 0 | 0
Libido increased (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Negative thoughts (Psychiatric disorders) | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 3 | 1 | 3
Sleep disorder (Psychiatric disorders) | 1 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 2 | 0 | 1
Proteinuria (Renal and urinary disorders) | 4 | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0
Balanitis (Reproductive system and breast disorders) | 2 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 5 | 1 | 2
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Perineal ulceration (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 2 | 0
Vaginal disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lymphadenectomy (Surgical and medical procedures) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hyperaemia (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1
Labile hypertension (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.